CLINICAL TRIAL: NCT02626208
Title: A Dose Finding Study to Evaluate Serum Estradiol Levels With Use of Contraceptive Vaginal Rings Releasing Nestorone® and Escalating Doses of Estradiol in Normal Cycling Women
Brief Title: Dose Finding Study of Contraceptive Vaginal Ring With Different Estradiol Levels in Combination With Nestorone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Population Council (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCN012A
Record Dates: First submitted 2015-11-10; First posted 2015-12-10 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Suppression of Ovulation
Keywords: Contraceptive vaginal ring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nestorone®/ Estradiol 75 (Experimental): Device: Nestorone®/Estradiol Contraceptive Vaginal Ring with 200 mcg/day of NES and 75 ug/day of estradiol
  Interventions: Device: Nestorone®/Estradiol Contraceptive Vaginal Ring
- Nestorone®/Estradiol 100 (Experimental): Device: Nestorone®/Estradiol Contraceptive Vaginal Ring with 200 mcg/day of NES and 100 ug/day of estradiol
  Interventions: Device: Nestorone®/Estradiol Contraceptive Vaginal Ring
- Nestorone®/ Estradiol 200 (Experimental): Device: Nestorone®/Estradiol Contraceptive Vaginal Ring with 200 mcg/day of NES and 200 ug/day of estradiol
  Interventions: Device: Nestorone®/Estradiol Contraceptive Vaginal Ring

INTERVENTIONS:
Device: Nestorone®/Estradiol Contraceptive Vaginal Ring — Three arms of contraceptive vaginal rings contain a fixed dose (200 mcg/day) of Nestorone® and escalating doses (75 µg/d, 100 µg/d, or 200 µg/d /day) of estradiol

SUMMARY:
This clinical trial investigates a new vaginal delivery system made of silicone rubber, containing Nestorone®, a 19-nor progesterone derivative and a low dose of serum estradiol (E2). The investigators plan to evaluate one-month data on the serum estradiol (E2) levels of three different contraceptive vaginal rings that contain a fixed dose of NES and escalating doses (75 µg/day, 100 µg/day, or 200 µg/day) of estradiol as the basis for selecting a CVR for a larger contraceptive efficacy trial.

DETAILED DESCRIPTION:
This dose-finding study aims to evaluate serum estradiol levels with use of contraceptive vaginal rings releasing Nestorone® and escalating doses of estradiol in normal cycling women. The primary objective is to evaluate one-month data on the serum estradiol (E2) levels of three different contraceptive vaginal rings containing a fixed dose of Nestorone® (NES) and escalating doses of estradiol as the basis for selecting a contraceptive vaginal ring (CVR) dose for a contraceptive efficacy trial. The secondary objectives are to evaluate the effects of three different estradiol doses of a NES- E2 CVR on progesterone levels, bleeding and side effects during one month of use and to evaluate the effects of a hormone-free internal on bleeding patterns. Nestorone serum levels will further be measured as an indication of compliance with the continuous use of the ring.

ELIGIBILITY:
Inclusion Criteria:

1. Good general overall health with no chronic medical conditions that result in periodic exacerbations that require significant medical care.
2. Age 18-39 years, inclusive, at the enrollment visit.
3. Have a regular menstrual cycle 21-35 days in duration when not using hormonal contraception
4. Have an intact uterus and both ovaries.
5. Able and willing to comply with the protocol and sign an informed consent.
6. Consistent use of effective contraception during the preceding cycle (note: women who use oral, transdermal, vaginal, implantable or intrauterine hormonal contraceptives in the preceding cycle must have discontinued at least 7 days prior to start of treatment and not had unprotected intercourse since discontinuing the method).
7. Not at high risk for pregnancy, defined as consistently using a non-hormonal method of contraception (including Copper IUDs); have a surgically sterile male partner with a vasectomy; be abstinent; or be in a same-sex relationship from the start of treatment through study exit (including recovery period).
8. Have a negative pregnancy test at the admission visit.
9. Have a diastolic blood pressure (BP) ≤85 mm Hg and systolic BP ≤135 mm Hg after 5 minutes rest in sitting position at the admission visit.
10. Willing to abstain from use of non-water based vaginal lubricant during the study.

Exclusion Criteria:

1. Participating in another clinical trial involving an investigational product within the last 30 days (prior to screening) or planning to participate in another clinical trial during this study.
2. Not living in the catchment area of the study site.
3. Known hypersensitivity to progestins or estrogen.
4. Contraindications to combined estrogen-progestin contraceptive use including:

   * Thrombophlebitis or thromboembolic disorders.
   * Past personal history of deep vein thrombophlebitis or thromboembolic disorders.
   * History of venous thrombosis or embolism in a first-degree relative <55 years of age suggesting familial defect in blood coagulation system.
   * History of thrombosis or embolism OR any other personal or family history which in the opinion of the investigator suggests increased risk.
   * History of stroke.
   * Known or suspected carcinoma of the breast.
   * Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia.
   * Undiagnosed abnormal genital bleeding.
   * Cholestatic jaundice of pregnancy or jaundice with prior hormonal contraceptive use.
   * Hepatic adenomas or carcinomas.
   * Known or suspected pregnancy.
   * Smoking in women who are 35 years and over or will be 35 years during the course of the trial; women <35 years who smoke 15 cigarettes or more per day must be evaluated by the investigator for inclusion based on risk factors that would increase their risk for cardiovascular disease (CVD) and thromboembolism, e.g. lipid levels, glucose level, BP, BMI, family history of CVD at a young age.
   * History of retinal vascular lesions, unexplained partial or complete loss of vision.
   * Headaches with focal neurological symptoms (e.g., migraines with auras).
5. Desire to become pregnant during the study.
6. Breastfeeding.
7. Undiagnosed vaginal discharge or vaginal lesions or abnormalities. Subjects diagnosed at screening with a Chlamydia or gonococcus infection may be included in the trial following treatment; partner treatment is also recommended. Subjects with vaginal infection (yeast, trichomonis, or bacterial vaginosis) may be enrolled after treatment. Investigators should make a determination if subjects are at high risk for reinfection, e.g. multiple sex partners, untreated partner, and whether such subjects can be included. In accordance with PI/medical designee assessment and local standards of practice, women with a history of genital herpes can be included if outbreaks are infrequent.
8. A known clinically significant Pap test abnormality, as managed by current local or national guidelines that will require treatment during study participation.
9. Known benign or malignant liver tumors; known active liver disease.
10. Invasive cancer (past history of any carcinoma or sarcoma, except non-melanoma skin cancer).
11. Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive.
12. Known or suspected current alcoholism or drug abuse.
13. Elevated serum fasting clinical chemistry values or complete blood count (CBC) values designated clinically significant by the investigator or medically qualified sub-investigator.
14. Uncontrolled thyroid disease.
15. Known impaired hypothalamic-pituitary-adrenal reserve.
16. Body mass index (BMI) >35.
17. Use of injectable contraceptives (e.g. cyclofem or depo-medroxyprogesterone acetate) during the 9 months prior to enrollment or no spontaneous menses since last injection.
18. Use of oral, transdermal, vaginal, implantable or intrauterine contraceptives within 7 days prior to start of the treatment cycle. (Copper IUD is allowable. Levonorgestrel releasing IUD is not allowed.) NOTE: Discontinuation of any of these methods must have been for personal reasons unrelated to the purpose of enrollment in this study.
19. Known hypersensitivity to silicone rubber.
20. History of toxic shock syndrome.
21. Cystoceles or rectoceles or other anatomical abnormality that would preclude use of a vaginal ring.
22. Planning to undergo major surgery during study participation.
23. Severe constipation.
24. Use of liver enzyme inducers or inhibitors on a regular basis.
25. Known HIV infection.
26. Bariatric surgery within the past year prior to enrollment. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in serum estradiol (E2) levels of three different contraceptive vaginal rings | Assessments will be taken before insertion of the study ring (Day 1); Day 4 or ; Twice weekly during study ring use (approximately Days 7 or 8, 11 or 12, 14 or 15, 18 or 19, 21 or 22, 25 or 26) and at removal of study ring (Day 28-30)

SECONDARY OUTCOMES:
Change in progesterone levels | Assessments will be taken before insertion of the study ring (Day 1); Day 4 or ; Twice weekly during study ring use (approximately Days 7 or 8, 11 or 12, 14 or 15, 18 or 19, 21 or 22, 25 or 26) and at removal of study ring (Day 28-30)
Vaginal bleeding- amount and frequency | Assessments will be taken before insertion of the study ring (Day 1); Day 4 or ; Twice weekly during study ring use (approximately Days 7 or 8, 11 or 12, 14 or 15, 18 or 19, 21 or 22, 25 or 26) and at removal of study ring (Day 28-30)
Adverse event | Assessments will be taken before insertion of the study ring (Day 1); Day 4 or ; Twice weekly during study ring use (approximately Days 7 or 8, 11 or 12, 14 or 15, 18 or 19, 21 or 22, 25 or 26) and at removal of study ring (Day 28-30)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Blithe, MD, Study Chair — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (7):
- United States (7):
  - University of California, Davis, Sacramento, California
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science Unit, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School (EVMS), Norfolk, Virginia

REFERENCES:
- See also: The National Institute on Child Health and Human Development (NICHD) supports research on male and female contraception and conducts clinical trials of new contraceptive drugs and devices. — https://www.nichd.nih.gov/research/supported/Pages/cctn.aspx